CLINICAL TRIAL: NCT04660513
Title: Obesity-Related Glycine Deficiency: Investigating a Long-standing Metabolic Paradox Using Bedside and Bench Approaches
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Baylor College of Medicine (Other); National University Health System, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: SGH-ENDO-GlycineTA-001
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Glycine Metabolism Disturbances; Insulin Resistance; Morbid Obesity; Oxidative Stress
Keywords: glycine; obesity; bariatric surgery; gluthathione
MeSH Terms: conditions — Insulin Resistance; Obesity, Morbid; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morbid obesity: BMI 32.5 kg/m2 and above
  Interventions: Procedure: Bariatric surgery
- Non-obese healthy controls: BMI below 25 kg/m2

INTERVENTIONS:
Procedure: Bariatric surgery — Subjects with morbid obesity underwent bariatric surgery
  Groups: Morbid obesity

SUMMARY:
Obesity, in addition to causing abnormal glucose and lipid metabolism, is also associated with altered plasma concentrations of multiple amino acids, including increased levels of branched-chain amino acids and decreased levels of glycine. The mechanisms and consequences of obesity- related glycine deficiency are unknown.

The overall aim of this project is to comprehensively study glycine metabolic pathways in morbid obesity using stable-isotope tracer techniques in human subjects and validating kinetic findings using a cell model of oxidative stress.

This will be a single-centre, observational study. 21 individuals with morbid obesity scheduled for bariatric surgery and 21 non-obese controls will be recruit. They will undergo different study visits and procedures and the human biological materials collected will be analysed for as per aims of the studies. We believe that the glycine metabolic pathways, possibly through the optimization of gluthathione (GSH) synthesis, may provide targets to develop novel therapeutic agents.

DETAILED DESCRIPTION:
Metabolic tracers: 1,2-[13C2]-Glycine, 1,2-[13C2]-Glycine, 2,3,3,-[2H3]-Serine and [2H5]-Phenylalanine will be infused for quantification of various pathways associated with glycine metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-65 years
2. BMI < 25 kg/m2 for non-obese controls or BMI ≥ 32.5 kg/m2 for obese subjects scheduled for bariatric surgery
3. Able to provide informed consent

Exclusion Criteria:

All subjects:

1. Weight > 150 kg
2. Renal impairment (estimated creatinine clearance estimated by Cockcroft-Gault Equation < 60 ml/min)
3. Haemoglobin concentration < 10 g/L
4. Serum alanine aminotransferase or aspartate aminotransferase above 2x upper limit of normal
5. Uncontrolled hypertension (BP > 180/110 mmHg)
6. Pregnancy
7. Nursing mothers
8. Significant cardiovascular disease (e.g. acute myocardial infarction, congestive cardiac failure, ischemic heart disease, atrial fibrillation, sick sinus syndrome, supraventricular tachycardia)
9. Previous stroke
10. Uncontrolled thyroid disease
11. Surgery requiring general anaesthesia within 4-weeks before enrolment
12. Psychiatric disorders requiring medication
13. Significant alcohol intake (> 1 unit per day for women and > 2 units per day for men)
14. Subcutaneous insulin injections
15. Systemic steroid usage (eg. prednisolone, hydrocortisone, cortisone, dexamethasone)
16. Cancer within the last 5-years (except squamous cell and basal cell cancer of the skin)
17. Any factors likely to limit adherence to study protocol (e.g. dementia; alcohol or substance abuse; history of unreliability in medication taking or appointment keeping; significant concerns about participation in the study from spouse, significant other or family members)

Non-obese controls 1. Known Diabetes Mellitus (diagnosed according to 2014 Ministry of Health Clinical Practice Guidelines for Diabetes Mellitus)

Obese subjects

1. HbA1C < 9%

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Non-obese controls from our healthy volunteer database will be invited to participate. Obese subjects attending the weight management clinics in the hospital will be referred to the study team by their attending physicians
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Glycine kinetic | Baseline for all subjects and 5-12 months after bariatric surgery for morbid obesity group
  Differences in glycine kinetic measurements between obese subjects and controls, and within obese subjects after bariatric surgery
Insulin sensitivity | Baseline for all subjects and 5-12 months after bariatric surgery for morbid obesity group
  Differences in insulin sensitivity between obese subjects and controls, and within obese subjects after bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan HC, Hsu JW, Tai ES, Chacko S, Kovalik JP, Jahoor F. The impact of obesity-associated glycine deficiency on the elimination of endogenous and exogenous metabolites via the glycine conjugation pathway. Front Endocrinol (Lausanne). 2024 Apr 3;15:1343738. doi: 10.3389/fendo.2024.1343738. eCollection 2024. PMID 38633754
- [Derived] Tan HC, Hsu JW, Tai ES, Chacko S, Wu V, Lee CF, Kovalik JP, Jahoor F. De Novo Glycine Synthesis Is Reduced in Adults With Morbid Obesity and Increases Following Bariatric Surgery. Front Endocrinol (Lausanne). 2022 Jun 9;13:900343. doi: 10.3389/fendo.2022.900343. eCollection 2022. PMID 35757406